CLINICAL TRIAL: NCT00741286
Title: Study for the Multi-Center Placebo-Controlled Double-Blind Clinical Trial for the Evaluation of the Effect of Cilostazol on Pulsatility Index of Transcranial Doppler in the Acute Lacunar Infarction Patients
Brief Title: Effect of Cilostazol in the Acute Lacunar Infarction Based on Pulsatility Index of Transcranial Doppler
Acronym: ECLIPse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inje University (Other)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Jae Hyeon Park, MD, PhD, Sanggye Paik Hospital, Inje University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECLIPse
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Results first posted 2011-09-05 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2010-08

CONDITIONS: Cerebral Infarction
Keywords: Cerebral infarction; Cilostazol; Aspirin; Transcranial Doppler; Pulsatile Index
MeSH Terms: conditions — Cerebral Infarction | interventions — Aspirin; Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asprin (100mg) plus placebo (Placebo Comparator): Asprin (100mg) plus placebo
  Interventions: Drug: Aspirin
- Asprin (100mg) plus cilostazol (200mg) (Active Comparator): Asprin (100mg) plus cilostazol (200mg)
  Interventions: Drug: cilostazol

INTERVENTIONS:
Drug: Aspirin — Asprin (100mg) plus placebo
  Arms: Asprin (100mg) plus placebo
Drug: cilostazol — Aspirin (100mg) plus cilostazol (200mg)
  Other Names: Pletaal
  Arms: Asprin (100mg) plus cilostazol (200mg)

SUMMARY:
RATIONALE:

* Elevation in pulsatility indices (PIs), measured by transcranial Doppler (TCD), has been postulated to reflect downstream increased vascular resistance caused by small-vessel disease (SVD).
* Small arterial vessels are a significant determinant of vascular resistance and PIs are elevated when SVD is present in the intracranial circulation.
* Cilostazol, a phosphodiesterase III inhibitor, has other non-antiplatelet effects, such as vasodilation and neuroprotective effect. It has been shown to be effective in the secondary prevention of stroke especially in the SVD and it may be related to the other non-antiplatelet effects of cilostazol.

OBJECTIVES:

* In this study, we aim to investigate whether cilostazol affects the changes of PIs in patients with acute lacunar infarction using serial TCDs.
* Our hypothesis is that cilostazol has other non-antiplatelet effects such as vasodilation effect and may decrease the vascular resistance in patients with acute lacunar infarction. Hence, cilostazol will decrease the PIs in patients with acute lacunar infarction.

DETAILED DESCRIPTION:
TREATMENTS:

* Cilostazol is an agent inhibiting platelet aggregation.
* A matching placebo of cilostazol is an inactive substance that looks similar to the active cilostazol tablet.

TREATMENT PLAN:

* There will be two treatment groups; one will receive cilostazol 200mg (100mg twice per day), the second matching placebo of cilostazol.
* These study drugs will be administered on top of aspirin (100mg) systematically prescribed to such patients

PRIMARY ENDPOINT:

* The changes of PI between the baseline and 14 and 90 days follow-up study.

STUDY EXECUTION:

* Two hundred sixty patients, presenting with first ever lacunar infarction within 7 days after the onset of symptoms will be recruited within two years.
* Patients will be followed up during the three months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first ever lacunar infarction within 7 days after the onset of symptoms
* Age: more than 45 years of age

Exclusion Criteria:

* Patients with any contraindications to the treatment with antiplatelet therapy
* Patients with potential cardiac embolic source; prosthetic valve, atrial fibrillation, atrial flutter, left atrial/atrial appendage thrombus, sick sinus syndrome, left ventricular thrombus, dilated cardiomyopathy, akinetic or hypokinetic left ventricular segment, atrial myxoma, Infective endocarditis, mitral valve stenosis or prolapse, mitral annuls calcification, left atrial turbulence, nonbacterial endocarditis, congestive heart failure, recent myocardial infarction (within 4 weeks)
* Bleeding diathesis
* Chronic liver disease (ALT > 100 or AST > 100) or chronic renal disease (creatinine > 3.0mg/dl)
* Anemia (hemoglobin < 10mg/dl) or thrombocytopenia (platelet count less than 100,000/mm3)
* Nonatherosclerotic vasculopathy; patients with clinical characteristics suggesting arterial dissection, moyamoya disease, Takayasu's arteritis, radiation associated angiopathy, and other vasculitis.
* Pregnant or lactating patients
* Patients with hyperthyroidism or COPD
* Patients with current anticoagulation or antiplatelet therapy
* Patients with poor temporal window in transcranial Doppler

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hyeon Park, MD, PhD, Principal Investigator — Sanggye Paik Hospital, Inje University College of Medicine
Locations (8):
- South Korea (8):
  - Sanbon Medical Center, Gunpo
  - National Health Insurance Corporation Ilsan Hospital, Ilsan
  - Bundang CHA Hospital, Seongnam
  - National medical center, Seoul
  - Yongdong Severance Hospital, Seoul
  - Sanggye Paik Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Wonju Christian Hospital, Wŏnju

REFERENCES:
- [Derived] Han SW, Lee SS, Kim SH, Lee JH, Kim GS, Kim OJ, Koh IS, Lee JY, Suk SH, Lee SI, Nam HS, Kim WJ, Yong SW, Lee KY, Park JH. Effect of cilostazol in acute lacunar infarction based on pulsatility index of transcranial Doppler (ECLIPse): a multicenter, randomized, double-blind, placebo-controlled trial. Eur Neurol. 2013;69(1):33-40. doi: 10.1159/000338247. Epub 2012 Nov 1. PMID 23128968

RESULTS

PARTICIPANT FLOW:
Recruitment Details: ECLIPse was designed as a multicenter, randomized, double-blind, placebo-controlled trial. Between November 2006 and October 2008, 203 patients were consecutively enrolled from eight tertiary-care hospitals.
Pre-assignment Details: A total of 513 patients who had experienced their first classic lacunar syndromes were screened for study enrollment, of which 101 (19.7% of the screened population) refused to participate in the study. Seventy-four patients (14.4%) were not eligible for the trial, and 135 (26.3%) were excluded by the exclusion criteria.
Groups:
- Asprin Plus Placebo: Placebo twice a day on top of aspirin 100mg a day
- Asprin Plus Cilostazol: Cilostazol (100mg) twice a day on top of aspirin 100mg a day
Period: Overall Study
Arm/Group | Asprin Plus Placebo | Asprin Plus Cilostazol
Started | 103 | 100
Completed | 83 | 81
Not Completed | 20 | 19
Not completed — Lost to Follow-up | 15 | 10
Not completed — Adverse Event | 1 | 6
Not completed — Protocol Violation | 3 | 2
Not completed — Primary Outcome | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asprin Plus Placebo | Asprin Plus Cilostazol | Total
Number analyzed (Participants) | 103 | 100 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 45 | 92
  >=65 years | 56 | 55 | 111
Age Continuous [Mean (Standard Deviation); unit: years] | 65.48 (9.92) | 64.63 (9.07) | 65.06 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 78 | 74 | 152
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 103 | 100 | 203

OUTCOME MEASURES:

1. Primary Outcome: The Changes of Middle Cerebral Artery (MCA) and Basilar Artery (BA) Pulsatility Index (PI) at 14 and 90 Days From the Baseline Transcranial Doppler (TCD) Study
Description: The PI is designed to measure vascular resistance and characterizes the shape of the spectral waveform. For the study, the mean, systolic, and diastolic flow velocities were measured using TCD. Gosling's PI was determined as the difference between the peak systolic and end-diastolic velocities divided by the mean flow velocity in each artery.The changes of MCA and BA PIs at 14 and 90 days from the baseline TCD study was calculated for the study.
Time Frame: 14 days and 90 days from the baseline TCD study
Population: Of the 203 patients included in the intention-to-treat analysis, 164 were included in the per-protocol analysis of the primary outcome.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Asprin Plus Placebo | Asprin Plus Cilostazol
Number analyzed (Participants) | 83 | 81
ratio
  Changes of PI in Right MCA (14 days) | 0.07 (0.13) | 0.08 (0.13)
  Changes of PI in Right MCA (90 days) | 0.09 (0.13) | 0.14 (0.13)
  Changes of PI in Left MCA (14 days) | 0.08 (0.13) | 0.1 (0.14)
  Changes of PI in Left MCA (90 days) | 0.07 (0.13) | 0.13 (0.13)
  Changes of PI in BA (14 days) | 0.09 (0.14) | 0.09 (0.14)
  Changes of PI in BA (90 days) | 0.1 (0.18) | 0.18 (0.16)
Statistical Analysis 1: Comparison: Asprin Plus Placebo vs Asprin Plus Cilostazol; A linear mixed model for a repeated measures covariance pattern model with unstructured covariances within subjects was used. Two fixed effects were included: 1 between-subjects treatment effect (group: cilostazol, control) and 1 within-subject time effect (time: baseline, 14 days, 90 days). A possible difference in treatment across 14- and 90-day follow-up was analyzed by time x treatment interactions; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: Asprin Plus Placebo vs Asprin Plus Cilostazol; To determine between-group differences of changes in the PIs at 14 and 90 days from the baseline study; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Number of Patients With First Recurrent Stroke of Any Type
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | Asprin Plus Placebo | Asprin Plus Cilostazol
Number analyzed (Participants) | 83 | 81
participants | 1 | 1
Statistical Analysis 1: Comparison: Asprin Plus Placebo vs Asprin Plus Cilostazol; Test type: Superiority or Other; p < 0.05, Chi-squared

ADVERSE EVENTS:
Arm/Group | Asprin Plus Placebo | Asprin Plus Cilostazol
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/81
Other Adverse Events (participants affected / at risk) | 0/103 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No